CLINICAL TRIAL: NCT04085432
Title: Validation Study for a Frailty Self Assessment Tool in Retirees Aged 70 and Over
Brief Title: Validation of a Frailty Self Assessment Tool
Status: Completed | Type: Observational
Sponsor: International Longevity Centre France (Other)
Responsible Party: Sponsor
Other Study IDs: CNAV- ILC France 2; 2018-A03324-51 (Other: ANSM)
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Self administered questionnaire and Clinical evaluation — Self administered questionnaire and clinical evaluation

SUMMARY:
The number of elderly is increasing throughout of the world. Aging is associated with increasing diseases that may be preventable. Over the last decades, frailty has emerged as one of the major risk factors for loss of autonomy. Frailty can be reversed through appropriate interventions particularly when they are implemented early. Therefore, early detection of frailty is a major objective. The goal of this study is to identify elderly subjects aged 70 years and over at the early stage of frailty by using a self administered questionnaire sent to the participant by mail. The results of the self assessment will be compared to the Fried criteria collected by a clinical examination conducted by a healthcare Professional blinded to the self assessment results.

DETAILED DESCRIPTION:
Five thousands (5000) retirees aged 70 and over will be randomly selected from National Retirement Pension Institute (CNAV) retirees (2500 living in Paris and 2500 living in Toulouse). They will receive a letter from the CNAV explaining the study approach and a separate self-assessment frailty questionnaire to be filled in by the retirees at home and sent back in a pre-paid envelope to International Longevity Centre France (ILC-France).

Retirees who have accepted the home assessment are examined by a healthcare professional, blinded to the results of self-administered questionnaire, using the Fried's frailty criteria in order to confirm or infirm the diagnosis of frailty.

The General practitioner will be informed of the investigation results in order to set up a personalized prevention plan.

ILC-France will anonymize both the self-administered questionnaires and the Fried assessments and send them to the Mixed Research Unit (UMR) 1027 in Toulouse.

Comparison of the Fried assessment results with those of the self-questionnaire will confirm the metrological characteristics (false negative, false positive, sensitivity, specificity, predictive value) of the questionnaire.

Secondary analyses will be conducted to compare the prevalence of frailty by age and gender.

The statistical analysis is carried out by the UMR 1027 of Toulouse.

ELIGIBILITY:
Inclusion Criteria:

* Retirees from the National Old-Age Insurance Fund
* Aged 70 or older,
* Living at home
* Representatives of the general population

Exclusion Criteria:

* Institutionalized retirees
* Retirees receiving the Personalised Allowance for Autonomy
* Retirees who enrolled in previous studies

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Retirees aged 70 and over, living at home
Sampling Method: Probability Sample
Enrollment: 5134 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Frailty and pre-frailty diagnosis rate | October 2019 to August 2020
  Frailty and pre-frailty diagnosis rate are detected by self administered questionnaire and confirmed by the Fried's frailty phenotype assessment

SECONDARY OUTCOMES:
Prevalence of frailty by age and gender | October 2019 to August 2020
  Prevalence of frailty by age and gender

CONTACTS AND LOCATIONS:
Overall Officials: Françoise FORETTE, MD, Principal Investigator — ILC France and Universite Paris Descartes
Locations (2):
- France (2):
  - Broca Hospital Geriatric Department, Paris
  - GERONTOPOLE of the Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided